CLINICAL TRIAL: NCT07242183
Title: Acute Effects of Hot-pack Therapy on Lumbar Erector Spinae Muscle Stiffness and Pain in Adults With Low Back Pain: A Randomised Controlled Trial.
Brief Title: Acute Effects of Hot-Pack Therapy in Low Back Pain
Acronym: HOTPACK-LBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Collaborators: Amasya University (Other); Ataturk University (Other)
Responsible Party: Principal Investigator, esedullah akaras, Dr., Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETU-PMR-HOTPACK-2025-RCT-v3
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Low Back Pain; Back Pain
Keywords: Hot-pack; Muscle Stiffness; Erector Spinae; Myotonometry
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Hyperthermia, Induced; Diathermy

STUDY DESIGN:
Intervention Model Description: Two-arm, single-session randomized controlled trial comparing moist hot-pack versus sham (room-temperature pack) in adults with nonspecific low back pain. Participants are randomized 1:1; treating therapist is not blinded, while participants and outcomes assessors are blinded. Outcomes: pain (VAS) and lumbar erector spinae stiffness (MyotonPro) immediately post-session; ODI at 24-48 h.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants receive either a heated moist pack or an identical setup with a room-temperature pack; identical towel barriers and procedures maintain participant blinding. The treating therapist cannot be blinded due to the nature of heat delivery. Outcome assessors are blinded to allocation; data are recorded with coded IDs to preserve blinding during analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot-Pack Therapy (Experimental): Single-session moist hot-pack applied to the lumbar region. Pack surface temperature ≈60-65 °C; 6-8 towel layers as barrier; total duration 20 minutes. Skin checks at minutes 5 and 10. Outcomes: pain (VAS) and erector spinae stiffness (MyotonPro) immediately post-session; ODI at 24-48 h
  Interventions: Device: Hot-Pack; Device: Sham Pack
- Room-Temperature Pack (Sham) (Sham Comparator): Single-session room-temperature pack applied to the lumbar region using the same setup as the active arm (identical towels/barrier, positioning, and timing) but without heat. Total duration 20 minutes. Outcomes measured on the same schedule. Maintains participant and assessor blinding.
  Interventions: Device: Hot-Pack; Device: Sham Pack

INTERVENTIONS:
Device: Hot-Pack — Thermal therapy delivered via a moist hot-pack applied to the lumbar area for 20 minutes. Target pack surface temp ≈60-65 °C at application; 6-8 towel layers to prevent burns; patient positioned prone or side-lying per comfort. Skin integrity checked at minutes 5 and 10; session stopped if adverse reactions occur. Single session only.
  Other Names: Thermotherapy; Heat therapy
Device: Sham Pack — Placebo thermotherapy control using a room-temperature pack with identical preparation, towel barriers, positioning, and duration (20 minutes) as the active intervention. No heat is delivered. Used to preserve participant blinding.
  Other Names: Placebo thermotherapy; Room-temperature pack

SUMMARY:
This single-centre, parallel-group randomized controlled trial will test whether one session of moist hot-pack therapy produces immediate improvements in pain intensity and lumbar erector spinae muscle stiffness in adults with nonspecific low back pain. Participants are randomized 1:1 to hot-pack or sham (room-temperature pack). Outcomes are assessed at baseline and immediately after the session using VAS (0-10 cm) and MyotonPro; a short follow-up (24-48 h) captures Oswestry Disability Index (ODI) and perceived change. The intervention is brief, low-risk, and commonly used in clinical practice, yet high-quality evidence on its acute effects is limited.

DETAILED DESCRIPTION:
Rationale. Hot-pack (thermotherapy) is frequently prescribed to reduce pain and muscle tension in low back pain, but controlled evidence quantifying immediate changes in muscle mechanical properties and pain remains scarce. Demonstrating short-term benefits with objective measures (MyotonPro) and validated scales (VAS, ODI) could inform pragmatic care pathways for nonspecific low back pain.

Objectives and Hypotheses. Primary objective: determine whether a single hot-pack session reduces erector spinae stiffness (MyotonPro) and pain (VAS) versus sham. Secondary objective: explore short-term effects on functional disability (ODI) and perceived improvement. We hypothesize greater immediate reductions in stiffness and pain, and better short-term function, with hot-pack versus sham.

Design and Setting. Prospective, two-arm, parallel RCT at Atatürk University Faculty of Medicine (Physical Medicine & Rehabilitation / Orthopedics). Target sample: 30 adults (pilot). Allocation is 1:1 using computer-generated randomization; outcome assessors and participants are blinded.

Participants. Adults 18-65 y with nonspecific/mechanical low back pain and baseline VAS ≥ 3/10. Key exclusions include pregnancy, pacemaker/implanted devices, recent lumbar surgery or heat/cold therapy (<6 weeks), dermatologic lesions, neurologic deficit, tumour, or systemic inflammatory disease. Written informed consent is obtained before any procedure.

Interventions.

Hot-pack (Active): Moist hot-pack at 60-65 °C applied over the lumbar region for 20 minutes with a 6-8 towel barrier. Skin is checked at minutes 5 and 10.

Sham (Comparator): Identical setup using a room-temperature pack (no heat).

Outcome Measures and Timing.

Primary: Change in pain intensity (VAS, 0-10 cm) from pre- to immediate post-intervention.

Key Secondary: Change in erector spinae stiffness (MyotonPro) from pre- to immediate post-intervention; ODI at 24-48 h; patient-reported perceived change.

Procedures. After screening and consent, baseline demographics and outcomes are recorded. MyotonPro measurements are taken over the lumbar erector spinae at L3-L4, 2-3 cm lateral, with three repeats per point and averaged. Post-session, VAS and MyotonPro are repeated; ODI and a brief perceived-change item are collected 24-48 h later. All assessments are performed by trained physiotherapists following device protocols and the Declaration of Helsinki.

Randomization, Masking, and Data Handling. Randomization is computer-assisted (1:1). Participants and assessors are blinded to group assignment via a sham procedure mirroring the active setup. Data are recorded with coded IDs and analysed with mixed-model repeated-measures ANOVA (group × time), reporting effect sizes and 95% CIs.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years

Nonspecific/mechanical low back pain (clinical diagnosis)

Baseline pain ≥3/10 on a 0-10 Visual Analogue Scale (VAS)

Able to understand procedures and provide written informed consent

Able to attend baseline, immediate post-session, and 24-48 h follow-up assessments

Exclusion Criteria:

* Neurologic deficit, tumour, or systemic inflammatory disease

Prior lumbar spine surgery

Heat or cold therapy to the lumbar region within the past 6 weeks

Dermatologic lesions, open wounds, or skin conditions over the lumbar area

Contraindications to heat (e.g., impaired sensation/neuropathy over the area, severe circulatory disorders)

Pregnancy

Implanted electronic devices (e.g., pacemaker)

Inability to comply with the study schedule or procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Lumbar Erector Spinae Stiffness (MyotonPro, N/m) From Baseline to Immediate Post-Intervention | Baseline and immediately post-session (~20-30 minutes)
  Myotonometric stiffness (N/m) is captured over lumbar erector spinae (L3-L4 level, ~2-3 cm lateral). Three taps per point; averaged. Endpoint is change score (Post - Baseline); negative values indicate reduced stiffness.

SECONDARY OUTCOMES:
Change in Pain Intensity (VAS, 0-10) From Baseline to Immediate Post-Intervention | Baseline (pre-session) and immediately post-session (~20-30 minutes after start
  Pain intensity is measured on a 10-cm Visual Analogue Scale (0=no pain, 10=worst pain). The primary endpoint is the change score (Post - Baseline); negative values indicate improvement. Participants rate pain just before the session and immediately after the 20-minute intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan YAĞIZ, Dr., Study Chair — Amasya University; Julian OWEN, Dr., Study Director — Bangor University

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data. Only aggregate findings will be reported in publications and at ClinicalTrials.gov.